CLINICAL TRIAL: NCT04697706
Title: Effect of a High Citrate Beverage on Urine Chemistry in Urinary Stone Disease
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-01153
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Urinary Stone
MeSH Terms: conditions — Urinary Calculi | interventions — Water

STUDY DESIGN:
Intervention Model Description: All participants will undergo the same two study periods. The order of the periods will be randomly assigned to each patient in order to eliminate the possibility of a sequence effect. The study periods can be done in non-consecutive weeks, chosen at the patients' discretion. The periods will each be 1 week in duration.
Masking Description: Given the nature of the two arms, it is not possible to blind the participants or investigators.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study period "Water" (Active Comparator): Participants will take in 1L of tap water per day plus ad lib, self-selected fluids.
  Interventions: Other: Water
- Study period "Moonstone" (Experimental): Participants will take one packet of Moonstone powder reconstituted in 500 ml water, twice a day, to total 1 L per day (66 meq of potential alkali/day) plus ad lib fluids. Moonstone packets will be supplied by Dr. Arnie's, Inc.
  Interventions: Dietary Supplement: Moonstone

INTERVENTIONS:
Dietary Supplement: Moonstone — Participants will take one packet of Moonstone powder reconstituted in 500 ml water, twice a day, to total 1 L per day (66 meq of potential alkali/day) plus ad lib fluids. Moonstone packets will be supplied by Dr. Arnie's, Inc.
  Participants will follow their own self-chosen ad lib diets and complete a diet diary (Appendix) for days 6 and 7 in the first study period. On day 7, a 24-hour urine collection will be performed, and a 50-ml aliquot of urine will be sent to Litholink (Chicago, IL) via FedEx for analysis. Participants will then continue to the second study period and will use the diet diary completed in the first study period on days 6 and 7 to reproduce the identical diets for days 6 and 7 of the subsequent collection period.
  Arms: Study period "Moonstone"
Other: Water — Participants will take in 1L of tap water per day plus ad lib, self-selected fluids.
  Participants will follow their own self-chosen ad lib diets and complete a diet diary (Appendix) for days 6 and 7 in the first study period. On day 7, a 24-hour urine collection will be performed, and a 50-ml aliquot of urine will be sent to Litholink (Chicago, IL) via FedEx for analysis. Participants will then continue to the second study period and will use the diet diary completed in the first study period on days 6 and 7 to reproduce the identical diets for days 6 and 7 of the subsequent collection period.
  Arms: Study period "Water"

SUMMARY:
This study will investigate the effect of a patented high citrate beverage on urine chemistry in patients with urinary stone disease (USD). It is a minimal risk study of an over-the-counter beverage called Moonstone, which is commercially available. This study is considered preparatory for the RO-1 and is not intended to produce a definitive outcome regarding kidney stones.

ELIGIBILITY:
Inclusion Criteria:

The study will enroll patients with calcium, cystine and uric acid stone composition. Patients will be at least 18 years of age, with no upper limit of age. Patients will sign an informed consent form (ICF). We will seek participants who have experienced any USD events including renal colic with spontaneous stone passage, emergency room visits, or urological interventions, in the previous 5 years in order to encourage enrollment and adherence to the protocol. We will include all racial and ethnic groups, and both men and women. Besides stone composition, standard demographic data including gender, age, and body mass index will be collected.

Patients who are taking alkalinizing medications for prevention of USD including KCit, potassium bicarbonate, sodium citrate and sodium bicarbonate will be eligible for participation in the study. The patient's usual dose, however, will be discontinued for the 2 weeks which make up the two study periods. This maneuver will not be an important risk for stones for several reasons: 1) the period off alkali altogether will be one week; 2) the one week of Moonstone will offer a significant amount of alkali, likely as much or more than the patients' usual prescription doses; 3) participants will continue to adhere to fluid intake and dietary prescriptions.

These data are intended to be included in an RO-1 resubmission due November 5. We will therefore aspire to include 10 patients with calcium stones, 3 patients with cystine stones and 3 patients with uric acid stones.

Exclusion Criteria:

Investigators will exclude patients taking thiazides (indapamide, hydrochlorothiazide, and chlorthalidone). Our reasoning is that most calcium stone patients are not taking thiazides and such patients may be total body potassium-depleted (not necessarily reflected by serum potassium. Potassium depletion reduces citrate excretion (through effects on intracellular pH in the proximal tubule) so that patients taking thiazides could start with lower urine citrate excretion and have less of an increment in the Moonstone periods. The order of the periods might affect the magnitude of urine chemistry changes in those two periods.

Patients with chronic kidney disease tend to have reduced urinary citrate excretion due to mild metabolic acidosis. We will therefore exclude patients with estimated glomerular filtration rates (eGFRs) less than 60 ml/min/1.73 m2 calculated by the CKD-EPI equation. eGFRs will have been measured in the preceding year at a time when urinary tract obstruction due to USD was not present. We will also exclude women who are pregnant or nursing and people with any medical, psychiatric, debilitating disease/disorder, or social condition that in the judgment of the investigator would interfere with or serve as a contraindication to adherence to the study protocol or ability to give informed consent, or affect the overall prognosis of the patient.

The study will also exclude patients with a previous history of gastrointestinal intolerance, or any other intolerance of alkalinizing preparations. The proportion of USD patients who do not tolerate KCit is not clear. The Cochrane review on this topic states that there are adverse events reported with citrate therapy, but the effect was not statistically significant, in part because of incomplete reporting. Based on our experience, we usually cite this problem to affect about 10% of stone formers, with older people more frequently affected. We therefore do not think this exclusion criterion will have a sizable effect on enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2020-12-14 (Actual)

PRIMARY OUTCOMES:
Urine citrate excretion | 24 hours
  In calcium stone formers, the effect of Moonstone on urine citrate excretion will be compared to that of water in a non-inferiority analysis.
24-hour urine volume | 24 hours
  The effects of Moonstone on 24-hour urine volume, calcium excretion and SS will be compared.
24-hour urine pH | 24 hours
  The effect of Moonstone on 24-hour urine pH will be compared to that of water in a non-inferiority analysis in both cystine and uric acid stone formers
Increase in 24-hour urine citrate excretion | 24 hours
  A secondary outcome is an increase in 24-hour urine citrate excretion after Moonstone, compared with a period of water, in calcium stone-forming individuals.

CONTACTS AND LOCATIONS:
Overall Officials: David Goldfarb, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to the PI. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: beginning 9 months and ending 36 months following article publication
Access Criteria: Requests may be directed to the PI.